CLINICAL TRIAL: NCT04953481
Title: Home Care Needs and Current Nursing Status of Patients With Amyotrophic Lateral Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021023
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amyotrophic lateral sclerosis group: Patients with amyotrophic lateral sclerosis undergoing home care.
  Interventions: Other: survey
- Caregiver group: Caregivers

INTERVENTIONS:
Other: survey — The general information, home care status and functional status of ALS patients and family caregivers were collected.
  Groups: Amyotrophic lateral sclerosis group

SUMMARY:
The purpose of this study is to comprehensively investigate and analyze the home care needs and status quo of ALS patients in China, and to clarify their home care needs and status quo, so as to provide reference for the development of home care service planning and policy measures for ALS patients.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is the most common type of motor neuron disease. It is common in middle-aged and elderly people. Progressive skeletal muscle weakness, atrophy, fascicular fibrillation, bulbar paralysis and pyramidal tract sign are the main clinical manifestations. The survival time is usually 3-5 years. As the pathogenesis of ALS is not fully understood, there is no specific treatment for ALS. The clinical treatment mode of most patients with ALS is hospitalization at the end of the disease and maintenance treatment at home during the disease progression. At present, there are few reports on the home care needs and nursing status of ALS patients in China. This study is a cross-sectional survey. Based on consulting the relevant literature and consulting experts' opinions, the researchers designed the questionnaire of home care needs and nursing status of ALS patients, The convenience sampling method was used to select 126-252 ALS outpatients, 126-252 ALS inpatients, and 126-252 ALS family members from a third class a general hospital in Beijing. The needs and status of home care of ALS patients in China were comprehensively investigated and analyzed, and the needs and status of home care were clarified, so as to provide reference for the development of home care service planning and policy measures for ALS patients.

ELIGIBILITY:
Inclusion Criteria:

-

The inclusion criteria of ALS patients:

1. They met the diagnostic criteria of Chinese guidelines for the diagnosis and treatment of amyotrophic lateral sclerosis; ② Receiving care at home; ③ No cognitive impairment (if the patient is unable to talk and write due to illness, the family members can express it for the patient);

   ④ Informed consent, willing to participate in this study;

   ⑤ No mental illness.

   The inclusion criteria of caregivers: ① the primary caregiver designated by the patient was responsible for the primary care;
   * They are relatives of patients;

     * No payment for care; ④ Informed consent, willing to participate in this study;

       * No mental illness; ⑥ There was no cognitive impairment.

   Exclusion Criteria:

   -

   Exclusion criteria of ALS patients:

   ① severe physical diseases, such as malignant tumor, liver and kidney dysfunction, etc;

   ② They are participating in other intervention projects.

   Exclusion criteria of caregivers:
   * severe physical diseases, such as malignant tumor, liver and kidney dysfunction, etc; ② They are participating in other intervention projects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The outpatients, inpatients, discharged patients and their caregivers of ALS in a general hospital in Beijing.
Sampling Method: Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the Barthel index of ADL | At the time of survey (day 0)
  the Barthel index of ADL

SECONDARY OUTCOMES:
Caregiver Burden Inventory, CBI | At the time of survey (day 0)
  Caregiver Burden Inventory, CBI

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No